CLINICAL TRIAL: NCT05955703
Title: Evaluation of the Effect of the Training Program Based on the Precede-Proceed Model on Adherence to Treatment and Healthy Lifestyle Behaviors of Hemodialysis Patients
Brief Title: Evaluation of the Effect of the Training Program Based on the Precede-Proceed Model on Guality Life Style
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayşenur SARIASLAN, Assist. Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AYSENUR-TEZ
Record Dates: First submitted 2023-06-01; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Hemodialysis Patient
Keywords: Adherence to treatment; healthy lifestyle behavior; hemodialysis; nursing; precede-proceed model; quality of life
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using the experimental group as a result of the training based on PPM (Experimental): The training sessions planned within the scope of PPM were applied to the patients, who were divided into groups of six according to the bed order, for 15-20 minutes for eight weeks, when the patients felt well, through training booklets and power point presentations. When the trainings started, the posters prepared were hung in the waiting room while the intervention group was undergoing hemodialysis. The person providing the care of the patient was included in each training. During the trainings, it was requested that the training booklets be with the patients and the power point presentations continued in parallel with the training booklets.
  * Post-test was applied to intervention group
  * three months after the post-test application, follow-up test was applied to the intervention group in order to evaluate the impact.
  Interventions: Behavioral: ppm based training
- Using the control group as a result of the training based on PPM (No Intervention): After the follow-up test, training was given to the patients in the control group and a model-based training booklet was distributed.

INTERVENTIONS:
Behavioral: ppm based training — The training program based on the precede proceed model was applied to hemodialysis patients for 8 sessions. Eight sessions of training were given to the experimental group within the scope of the model, a booklet was developed in line with the trainings and posters were prepared.
  Arms: Using the experimental group as a result of the training based on PPM

SUMMARY:
This study was conducted to evaluate the effect of a Precede-Proceed Model-based (PPM-based) training program on treatment adherence, healthy lifestyle behaviors, and quality of life of hemodialysis patients.

DETAILED DESCRIPTION:
The Precede proceed model includes structured training phases to bring positive behavior change. The model, which consists of training phases, provides the researcher with the opportunity to identify the problem and the deficiencies that cause the problem, evaluate the quality of life with these deficiencies and develop a health program for its solution. In order to apply the nine-phase model, the individual-patient's voluntary cooperation, determination and active participation in health practices are required.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Hemodialysis treatment for at least 6 months,
* A total score of 1 or more from the Dialysis Diet and Fluid Restriction Non-Compliance Scale,
* A score between 1 and 7 on the scale of compliance with medical treatment,
* Place, time, person orientation,
* Does not have a psychiatric illness or a problem that prevents written or verbal communication,

Exclusion Criteria:

* Diagnosed with psychiatric illness Individuals with a diagnosis of malignancy wanting to leave research
* Those who do not attend all of the trainings / do not want to continue
* Individuals whose general condition is deteriorated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Effect of the Training Program based on the Precede-Proceed Model on quality of life style of Hemodialysis Patients | six month
  The patients' quality of life was evaluated with the SF-12 Quality of Life scale. The scale consists of 12 items. There is no breakpoint. The higher the score obtained from the scale, the higher the quality of life.

SECONDARY OUTCOMES:
2. Evaluation of the Effects of the Continuation Test (follow-up test results 3 months after the post-test) and the Education Program Based on the Pre-Continuation Model on the Quality of Life of Hemodialysis Patients | three month
  The patients' quality of life was evaluated with the SF-12 Quality of Life scale. The scale consists of 12 items. There is no breakpoint. The higher the score obtained from the scale, the higher the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)